CLINICAL TRIAL: NCT00752921
Title: Randomized Placebo Controlled Trial With Etoricoxib That is Taken to Prevent the Yom Kippur Headache
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shaare Zedek Medical Center (Other)
Responsible Party: Zev Wimpfheimer MD, Shaare Zedek Medical Center, Jerusalem Israel
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 54661.ctil
Record Dates: First submitted 2008-09-15; First posted 2008-09-16 (Estimated); Last update posted 2008-09-16 (Estimated); Status verified 2008-09

CONDITIONS: Headache
Keywords: Etoricoxib, Fasting Headache, Headache, Yom Kippur
MeSH Terms: conditions — Headache | interventions — Etoricoxib

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Active Comparator): Healthy Patients, age 18-65, who typically suffer from a Headache while fasting
  Interventions: Drug: etoricoxib
- B (Placebo Comparator): Healthy Patients, age 18-65, who typically suffer from a Headache while fasting
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: etoricoxib — 120 mg
  Arms: A
Drug: placebo — placebo
  Arms: B

SUMMARY:
Headache during fasting is a known entity in the scientific literature. The prevalence of such a headache is high and in a study conducted in Israel was found in 60% of people with a previous predilection for headache. A prior study showed a significant decrease in the incidence of fasting headache using rofecoxib, but the drug has been taken off the market. The goal of this project is to evaluate the efficacy of etoricoxib as treatment taken before the fast- a COX-2 inhibitor with a relatively long half life to prevent fasting induced headache. The study will be a prospective double blind placebo controlled trial using adult volunteers with a history of a fasting headache who will be abstaining from food and drink on Yom Kippur.

The study hypothesis is that treatment with etoricoxib prior to a 25 hour fast will decrease the incidence of fasting headache.

DETAILED DESCRIPTION:
Fasting is a known trigger for headache. More specifically, headache associated with ritual fasting in compliance with religious edict has been documented and described in the literature. These have been described in Jewish and Muslim ritual fasts, and have been dubbed 'Yom Kippur headache,' and 'First of Ramadan headache' respectively. The incidence of fasting associated headache during the 25 hour fast of Yom Kippur (YK) wherein no food or drink is ingested, has been documented in approximately 40% of participants, but as high as 66% of those prone to headache. (1) A recent study was published in which the authors were able to show a marked reduction in YK headache using rofecoxib 50mg, a Cox 2 specific nonsteroidal anti-inflammatory medication with a relatively long (17 hour) half life. In a placebo controlled double blind randomized trial, in a population with a history of fasting headache, the drug was ingested just prior to the start of the fast. The placebo group had an incidence of headache 65% of the time whereas the treatment group had an incidence of 19%. Headache in the treatment set was also on average milder than in the controls. These results were all significant statistically. (3)

Unfortunately for sufferers of fasting headache, rofecoxib (Vioxx), has been removed from the market and is no longer available.

We therefore propose to conduct a second study using etoricoxib (Arcoxia) - a Cox 2 specific antiinflammatory medication with a longer half life than rofecoxib.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 -65.
* Patients will be enrolled if they declared that they intended to complete the 25 hour YK fast, and had demonstrated their commitment by doing so for the previous three years (unless medically prevented.)
* We will only enroll patients who stated that they typically suffered from headache during the fast.

Exclusion Criteria:

* Patients with chronic medical problems including:

  * Heart disease,
  * Kidney disease,
  * Liver disease,
  * Peptic ulcer disease,
  * Hypertension,
  * Diabetes,
  * Lung disease including asthma,
  * History of gastrointestinal bleeding,
  * Patients with allergies or intolerance in the past to NSAIDs,
  * Pregnancy or lactation.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2008-09; Primary Completion 2008-10 (Estimated); Study Completion 2008-10 (Estimated)

PRIMARY OUTCOMES:
Incidence of Fasting Headache | 25 hours after administration

CONTACTS AND LOCATIONS:
Overall Officials: Zev S Wimpfheimer, MD, Principal Investigator — Shaare Zedek Medical Center, Jerusalem Israel
Locations (1):
- Shaare Zedek Medical Center, Jerusalem, Israel

REFERENCES:
- [Background] Drescher MJ, Elstein Y. Prophylactic COX 2 inhibitor: an end to the Yom Kippur headache. Headache. 2006 Nov-Dec;46(10):1487-91. doi: 10.1111/j.1526-4610.2006.00609.x. PMID 17115981
- [Background] Mosek A, Korczyn AD. Yom Kippur headache. Neurology. 1995 Nov;45(11):1953-5. doi: 10.1212/wnl.45.11.1953. PMID 7501139
- [Background] Awada A, al Jumah M. The first-of-Ramadan headache. Headache. 1999 Jul-Aug;39(7):490-3. doi: 10.1046/j.1526-4610.1999.3907490.x. PMID 11279933
- [Derived] Drescher MJ, Alpert EA, Zalut T, Torgovicky R, Wimpfheimer Z. Prophylactic etoricoxib is effective in preventing Yom Kippur headache: a placebo-controlled double-blind and randomized trial of prophylaxis for ritual fasting headache. Headache. 2010 Sep;50(8):1328-34. doi: 10.1111/j.1526-4610.2009.01587.x. Epub 2009 Dec 21. PMID 20039959